CLINICAL TRIAL: NCT00364091
Title: A Multi-Center, Randomized, Double-Masked Parallel Group Study Evaluating the Efficacy, Safety, and QOL of R89674 0.25% Ophthalmic Solution Compared to Vehicle or an Active Control in a Modified Model of Environmental Seasonal Allergic Conjunctivitis
Brief Title: Evaluation of Efficacy of Ophthalmic Solution in Seasonal Allergic Conjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vistakon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06-003-09
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Allergic Conjunctivitis
Keywords: allergic conjunctivitis, ophthalmology, multicenter, controlled
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Ophthalmic Solutions

INTERVENTIONS:
Drug: R89674 0.025% ophthalmic solution

SUMMARY:
The purpose of this summary is to evaluate the efficacy and safety of R89674 0.025% ophthalmic solution compared with placebo or an active control in subjects with seasonal allergic conjunctivitis

ELIGIBILITY:
Inclusion Criteria:

* history of positive diagnostic test for ragweed within the past 2 years;
* positive bilateral response to ragweed as induced by conjunctival allergen challenge

Exclusion Criteria:

* ocular infection;
* history of retinal detachment, diabetic neuropathy, or any progressive retinal disease;
* moderate to severe asthma;
* dry eye syndrome;
* history of severe, unstable, or uncontrolled cardiovascular, pulmonary, hepatic, renal or autoimmune disease;
* pregnancy or lactation

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2006-08; Primary Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Ocular itching and redness scores at defined timepoints

SECONDARY OUTCOMES:
QOL, severity of chemosis & redness, ocular itching and redness scores at defined timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Reza Haque, MD, Study Director — Vistakon Pharmaceuticals
Locations (6):
- United States (6):
  - Louisville, Kentucky
  - North Andover, Massachusetts
  - Creve Coeur, Missouri
  - Charlotte, North Carolina
  - Philadelphia, Pennsylvania
  - Memphis, Tennessee